CLINICAL TRIAL: NCT05965622
Title: Targeting Suicidality in Young Adults: a Randomized, Controlled Pragmatic, Multicentre Trial Evaluating the (Cost)-Effectiveness of Attachment Based Family Therapy Compared to Treatment as Usual
Brief Title: (Cost)-Effectiveness of ABFT for Suicidal Youth.
Acronym: REPAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: KU Leuven (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Principal Investigator, Claudi Bockting, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL82274.018.22; S65701 (Registry Identifier: REPAIR study)
Record Dates: First submitted 2023-07-07; First posted 2023-07-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Suicidal Ideation
Keywords: Suicidality in young adults; Attachment Based Family Therapy; (cost)-effectiveness
MeSH Terms: conditions — Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, pragmatic, multicentre, trial in the Netherlands and Belgium with 13 participating sites.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Part of the research team that will collect and analyse the data are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attachment Based Family Therapy + Treatment As Usual (Experimental): Attachment Based Family Therapy (ABFT) is a manualized treatment, that emerges from interpersonal theories that suggest suicide can be precipitated, exacerbated, or buffered against by the quality of family relationships. Parent(s)/caregiver(s) will be involved in the therapy.
  In the experimental group, patients will receive ABFT as an add-on therapy besides treatment as usual (TAU).
  Interventions: Behavioral: Attachment Based Family Therapy (ABFT) + Treatment As Usual (TAU)
- Treatment As Usual (Placebo Comparator): Treatment as Usual (TAU) contains all regular interventions that are currently used to treat suicidality. In the TAU group, a limited number of systemic family therapy sessions will be given (maximum 4 sessions).
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Attachment Based Family Therapy (ABFT) + Treatment As Usual (TAU) — Attachment Based Family Therapy (ABFT): ABFT is a manualized treatment, that emerges from interpersonal theories that suggest suicide can be precipitated, exacerbated, or buffered against by the quality of family relationships. Therefore, ABFT focuses on strengthening parent-child attachment bonds to create a protective and secure base for young adult development. Sessions are scheduled weekly, and the intervention lasts on average 16 weeks.
  The participants in the ABFT condition will also receive treatment as usual (TAU).
  Arms: Attachment Based Family Therapy + Treatment As Usual
Behavioral: Treatment As Usual (TAU) — The participants in the treatment as usual (TAU) condition will only receive regular existing care to treat suicidality in young adults.
  Arms: Treatment As Usual

SUMMARY:
Young adults who attempt to kill themselves is a common and serious mental health problem worldwide and certainly in Belgium and the Netherlands. Fatal suicide is the leading cause of death among young adults. It has devastating consequences both for the young adults themselves and for their families. It also has substantial economic costs. However, up until now, there is little research on the treatment of suicidality among young adults. The current psychological therapy approaches and drug treatments for young people at very high risk of fatal suicide attempts have only limited success. Increasing evidence indicates the importance of involving significant others in treatment and the importance of the unfulfilled need for belonging and secure attachment. The WHO recommends involving significant others in the treatment of suicidal young adults. However, in Belgium and the Netherlands, there is little knowledge on the effectiveness of family based treatments. Attachment Based Family Therapy, or ABFT, was shown to work well in several studies in the US. Also in Belgium and the Netherlands, ABFT is being used to treat suicidal young adults. However, how well it works compared to the current treatment and if it provides good value for money have not been studied in young adults. In the proposed study the investigators will test, in a real-life situation, whether ABFT works better than the current treatment and if it provides good value for money. This study is a collaboration between the Netherlands and Belgium and 6 or 7 sites will participate from each country. Sites can be hospitals, mental health centres, student health centres or private practices. Participants (138 individuals) are young adults between 18 and 25 years old who have frequent thoughts about killing themselves, and who seek mental health treatment. The investigators predict that, compared to current treatment, ABFT will reduce suicidal thoughts and suicide attempts and that this improvement will be maintained over time, and that it will be better value for money. The project will contribute to improving care for suicidal young adults with high suicide risk. Results will inform clinical guidelines and policymakers and improve the treatment of young adults with a high risk for fatal suicide, and their families.

DETAILED DESCRIPTION:
The investigators conduct a randomized controlled trial to evaluate the (cost-)effectiveness of ABFT compared to Treatment As Usual (TAU) on suicidality, as delivered in daily practice. The hypothesis is that, compared to TAU, ABFT will lead to a stronger reduction of suicidal ideation and suicidal behavior, and will be more cost-effective, will improve family functioning and young adult attachment, and that this effect will hold at follow-up. The primary objective is change in suicidality, that is, suicidal ideation, attempts and suicide as assessed by the Suicidal Ideation Questionnaire Junior (SIQ-JR), and as reported by therapists during treatment. Secondary objectives are cost-effectiveness, process, working alliance and adherence during treatment, and change in young adult depressive symptoms, family functioning, and young adult attachment.

Attachment Based Family Therapy (ABFT): ABFT is a manualized treatment, that emerges from interpersonal theories that suggest suicide can be precipitated, exacerbated, or buffered against by the quality of family relationships. Therefore, ABFT focuses on strengthening parent-child attachment bonds to create a protective and secure base for young adult development. Sessions are scheduled weekly, and the intervention lasts on average 16 weeks. Treatment as usual (TAU): Participants in both arms will receive TAU, in the experimental condition ABFT will be delivered as an add-on. Most treatment centres' clinical practices rely heavily on the use of antidepressants and/or CBT or DBT. All regular interventions are allowed in TAU, except for systemic family therapy of more than 4 sessions in total. Parents are allowed to be involved in the treatment, which is part of treatment as usual, and can comprise for instance psycho-education or parental support or skill training.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25.
* A score above 31 on the SIQ-JR (the cut-off for suicidality).
* Have at least one primary parent or caregiver that participates in the assessment and treatment. This could be a biological parent, stepparent, grandparent, other relative, or a foster parent.

Exclusion Criteria:

* Other DSM-5 disorders: substance dependency: severe alcohol or cannabis use disorder, all other substances: modest or severe substance use disorder.
* Severe conduct disorder.
* Evidence of psychotic features or prior psychosis (assessed with the SCID-5-S).
* Severe cognitive impairment (e.g., mental retardation, severe developmental disorders) as evidenced by educational records, parental report and/or clinical impression.
* Other circumstances that might affect participation (e.g., severe medical disorder, relocation).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Suicidality | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention, 12 months after intervention.
  Suicidality is assessed by the Suicide Ideation Questionnaire Junior (SIQ-JR; Reynolds & Mazza, 1999). Scores can range from 0 to 90, with a cut-off score of 31 indicating suicidality.

SECONDARY OUTCOMES:
Suicide ideation | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  Assessed with the SCID-5-S, the Structured Clinical Interview for DSM-5 Syndrome Disorders (Michael B. First, JBWW, Lorna Smith Benjamin, Robert L. Spitzer, 2017). The SCID-5-S is designed as a semi structured diagnostic interview for making the major DSM-5 diagnosis. Data obtained here are qualitative, f.i. 'Did you ever wish you were dead or that you would fall asleep and never wake up again? Can you tell me more about that?'.
Suicide attempts | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  Assessed with the SCID-5-S, the Structured Clinical Interview for DSM-5 Syndrome Disorders (Michael B. First, JBWW, Lorna Smith Benjamin, Robert L. Spitzer, 2017). The SCID-5-S is designed as a semi structured diagnostic interview for making the major DSM-5 diagnosis. Data obtained here are qualitative, f.i. 'did you ever try to kill yourself? If yes, what did you do? What happened then? Did you try to end your life?'.
Depression (DSM-5) | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  Assessed with the SCID-5-S, the Structured Clinical Interview for DSM-5 Syndrome Disorders (Michael B. First, JBWW, Lorna Smith Benjamin, Robert L. Spitzer, 2017). The SCID-5-S is designed as a semi structured diagnostic interview for making the major DSM-5 diagnosis. When 5 or more criteria are scored positive (from A1 - A9), there is an indication for a depressive disorder.
Depressive symptoms | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention, 12 months after intervention.
  Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001). With 0 = 'not at all' and 3 = 'nearly every day'. Scores of 1-4 = minimal depression, scores of 20-27 = severe depression.
Parental vision on the young adults depressive symptoms | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention, 12 months after intervention.
  Clinical Depression Inventory second edition (CDI-2; Bodden, Braet & Stikkelbroek, 2016). The CDI-2 for parents consists of 17 items, scored on a 4- point likert scale to indicate how often in the past 2 weeks symptoms occurred in their child. They respond to statements like "Looks sad" (0 not at all, 1 sometimes, 2 often, 3 almost always). A CDI-2 cut-off score of 16 is indicative of "significant" depressive symptoms according to the Dutch Mental Health Care guideline (Buitelaar et al., 2009: Multidisciplinaire Richtlijn GGZ, Addendum Depressie bij Jeugd, 2009).
Family functioning | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention, 12 months after intervention.
  Self-Report Measures of Family Functioning (SRFF; Stark et al., 1990), both the emerging adult and the parent(s)/caregiver(s). The SRFF is composed of 15 five-item factors (e.g., cohesion, conflict, and democratic family style). Items are Likert-type scales rated from 1 (very untrue) to 4 (very true). Items that are scored in reverse are: 2, 4, 5, 8 and 9. A higher score reflects better family functioning.
Attachment | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  To investigate whether ABFT improves young adult secure attachment, we will measure their Secure Base Script knowledge (i.e., implicit knowledge about how a care-related interaction unfolds, which participants only acquire if they are securely attached; Waters & Waters, 2006), using the Attachment Script Assessment (ASA; Waters & Waters, 2006; Waters et al., 2019; Waters & Roisman, 2019). The stories narrated by participants will be coded using a 7-point scale (higher scores reflect more SBS knowledge; H. S. Waters & Rodrigues-Doolabh, 2001). A score of 1 = no knowledge about a SBS, a score of 7 = a lot knowledge about a SBS.
Health-related quality of life | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  Health-related quality of life: 5 Level EQ-5D (EQ-5D-5L; Versteegh et al., 2016). The EuroQOL five dimensions (EQ-5D) is a short questionnaire used to assess utilities at each measurement. Utilities are converted into Quality-Adjusted Life Years (QALYs), using Dutch and Belgian tariffs. Scoring works as followed: for instance for the item 'Mobility', a score of 1 = 'I have no problems in walking about' and a score of 5 = 'I am unable to walk about'. Higher scores on the EQ-5D-5L reflect more perceived problems (i.e. perceived by the patient).
Disability | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0; Ustun, Kostanjsek, Chatterji & Rehm, 2010).
Non-suicidal self-injury | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention,12 months after intervention.
  Non-suicidal self-injury questionnaire (Buelens, Luyckx, Kiekens, Gandhi, Muehlenkamp & Claes, 2020). This is a self-report 5-item questionnaire that measures non-suicidal self-injury. Items reflect qualitative data of which non suicidal self injury behaviors someone has exhibited.
Autonomy | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention, 12 months after intervention.
  Autonomy of the young adult, as assessed by the questionnaire 'My Parents and I', a combination of items of the Emotional Autonomy Scale (EAS; Steinberg & Zilverberg, 1986) and the Psychological Separation Inventory (PSI; Hoffman 1984). Items are scored from 1 = 'not true at all' to 5 = 'totally true'. Some items (4, 6, 8, 13, 15) are scored in reverse. A higher score reflects less autonomy.
Entrapment | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 6 months after intervention, 12 months after intervention.
  Entrapment Short-Form Scale (E-SF; De Beurs et al., 2020). The E-SF is a 4-item questionnaire. Respondents are asked to indicate on a 5 point scale (0 = "not at all like me", 1 = "a bit like me", 2 = "moderately like me", 3 = "quite a bit like me", 4 = "extremely like me"), how much each statement applies to the respond. A higher score reflects a worse outcome (so a higher score reflects more entrapment feelings).
Health care and associated costs and costs from productivity loss | Measures change at: baseline, immediately after intervention, follow-up: 3 months after intervention, 12 months after intervention.
  Treatment Inventory of Costs in Patients with psychiatric disorders (TiC-P; Hakkaart-Van Roijen, 2002).

OTHER OUTCOMES:
Childhood Trauma | Baseline.
  Childhood Trauma Questionnaire (CTQ; Garnefski & Kraaij, 2001). This is a self-report 28-item questionnaire that measures 5 types of maltreatment: emotional, physical, and sexual abuse, and emotional and physical neglect. Items that are reverse coded, are: 2, 5, 7, 13, 19, 26, 28. Moderate-severe cutoff scores for each subscale are >= 13 for Emotional Abuse; >= 10 for Physical Abuse; >= 8 for Sexual Abuse; >= 15 for Emotional Neglect; and >= 10 for Physical Neglect.
Working Alliance Inventory | Every 2 months during intervention starting at the first session.
  Working Alliance Inventory (WAI; Horvath & Greenberg, 1986). Measures overall therapeutic alliance and consists of sub scales measuring (quality of therapy) tasks, goals and bonds. Administered to emerging adult and the participating parent(s)/caregiver(s). The total score of the WAI is calculated by adding up all of the items. Reverse items, 4, 8, 12, 16, are scored inversely: (5=1) (4=2) (2=4) (1=5). A higher score represents a stronger alliance.
Treatment fidelity | Every 2 months during intervention starting at the first session
  Treatment fidelity and non-verbal contact will be assessed via scoring the videotapes that ABFT therapists made of their sessions. This will be done by a trained researcher using the The Therapist Behavior Rating Scale-3 (TBRS-3; Diamond, Hogue, Diamond & Siqueland, 1996). Scores are given on a 6 point Likert-scale, with 0 = 'not at all' and 6 = 'thoroughly'. A higher score reflects a better outcome.
Therapy Procedure | Every 2 months during intervention starting at the first session
  Using the Therapy Procedure Checklist (TPC, Weersing, Wijs & Donenberg, 2002), which assesses therapists' reports of the techniques they employ when working with child and adolescent clients, and will be used to monitor Treatment as Usual in both study arms. TPC items encompass the 3 most common therapeutic models for youth: psychodynamic, cognitive, and behavioural.
Demographic characteristics and other parameters | Baseline
  Demographic characteristics: age, country of birth, current country, country of school, level of education, nationality, ethnicity, marital status, gender (or sex), ethnicity, level of education, gender identity (only applicable to young adults), medication use (only applicable to young adults), substance use (smoking, alcohol, drugs), gambling, psychiatric history (therapy, medication, number of previous episodes, duration of episodes and treatment), psychological help (current and past), number of siblings (only applicable to young adults), current family situation, number of children living at home (only applicable to parent(s)/caregiver(s)), relation to participant (only applicable to parent(s)/caregiver(s)), employment situation, work disability (if not employed), work disability benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia van der Spek, PhD, Study Director — Academic Medical Center (AMC); Claudi Bockting, professor, Principal Investigator — Academic Medical Center (AMC); Guy Bosmans, Professor, Study Director — KU Leuven
Locations (13):
- Belgium (6):
  - Prakijkt ConnectUs, Tongeren, Limburg
  - UGent Centrum Kind en Adolescent, Ghent, Oost-Vlaanderen
  - UPC KU Leuven, campus Kortenberg, Kortenberg, Vlaams-Brabant
  - PraxisP, Leuven, Vlaams-Brabant
  - STUVO Psychologen en Psychiaters, Leuven, Vlaams-Brabant
  - Praktijk Annemie Uyttersprot, Merchtem, Vlaams-Brabant
- Netherlands (7):
  - GGzE, Eindhoven, North Brabant
  - GGZ Oost Brabant, Oss, North Brabant
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Arkin, Amsterdam, North Holland
  - Levvel, Amsterdam, North Holland
  - Kenter Jeugdhulp, Santpoort-Noord, North Holland
  - GGz Centraal, Amersfoort, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bockting C, Bosmans G, Bergers N, Gavan L, Hiligsmann M, de Beurs D, Molenberghs G, Wijnen B, Lokkerbol J, van der Spek N. The effectiveness and cost-effectiveness of attachment-based family therapy for young adults with high suicidal ideation: protocol of a randomized controlled trial. Trials. 2024 Oct 16;25(1):686. doi: 10.1186/s13063-024-08499-7. PMID 39415182